CLINICAL TRIAL: NCT02824042
Title: An Open Label, Phase I Study to Assess the Effect of Itraconazole (CYP3A4 and P-gp Inhibitor) on the Pharmacokinetics of Anetumab Ravtansine and to Assess the ECG Effects, Safety and Immunogenicity of Anetumab Ravtansine Given as a Single Agent and Together With Itraconazole in Subjects With Mesothelin-expressing Advanced Solid Cancers
Brief Title: Thorough ECG (Electrocardiogram) and Drug Interaction Study With Anetumab Ravtansine and Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18329; 2017-001978-42 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Medical Oncology
Keywords: Phase 1; Solid tumors; Mesothelin; Itraconazole; PK DDI; ECG thorough QTC
MeSH Terms: interventions — anetumab ravtansine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anetumab ravtansine (Experimental): The evaluation of multiple ECG parameters and the drug-drug interaction (DDI) potential of anetumab ravtansine parameters when administered alone and together with itraconazole 100 mg oral capsules will be conducted in 2 sequential parts. On Cycle 1 Day 1, anetumab ravtansine will be given alone at a dose of 6.5 mg/kg in Part 1 and Part 2. On Cycle 2 Day 1, anetumab ravtansine will be given together with itraconazole at a dose of 0.6 mg/kg in Part 1, and at a dose of 6.5 mg/kg (planned) in Part 2.
  Interventions: Drug: Anetumab ravtansine (BAY94-9343); Drug: Itraconazole

INTERVENTIONS:
Drug: Anetumab ravtansine (BAY94-9343) — Anetumab ravtansine given IV On Day 1 of each 21-day treatment cycle Part 1: Cycle 1 Day 1: 6.5 mg/kg of body weight (BW) Cycle 2 Day 1: 0.6 mg/kg BW Part 2: Cycle 1 Day 1: 6.5 mg/kg BW Cycle 2 Day 1: 6.5 mg/kg BW (planned dose) Continuous treatment: Cycles ≥3 Day 1: 6.5 mg/kg BW once every 3 weeks (Q3W)
Drug: Itraconazole — Itraconazole 100 mg oral capsules given by mouth Cycle 1 (Day 18): 200 mg twice daily (BID) (Days 19 - 21): 200 mg once daily (QD) Cycle 2 (Days 1-8): 200 mg QD 12 days in total (Part 1 or Part 2)

SUMMARY:
Characterize the safety, tolerability, ECG effects, pharmacokinetics and immunogenicity of anetumab ravtansine given as single agent and after inhibition of CYP3A4 and P-gp by concomitant administration of itraconazole in subjects with mesothelin-expressing advanced solid cancers

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed, locally advanced or metastatic solid cancers of the following histological types:

  1. predominantly epithelial (≥50% tumor component) pleural or peritoneal mesothelioma
  2. epithelial ovarian cancer (fallopian tube and primary peritoneal cancers are eligible)
  3. adenocarcinoma of the pancreas,
  4. triple-negative adenocarcinoma of the breast
  5. non-small-cell adenocarcinoma of the lung
  6. gastric cancer (including gastro-esophageal junction)
  7. colon cancer
  8. cholangiocarcinoma
  9. Thymic carcinoma
* Subjects must have no standard therapy available, or have actively refused standard therapy
* Subjects must provide samples of archival tumor tissue collected and submitted anytime during the study
* Subjects must have a life expectancy of at least 12 weeks
* Subjects must have ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* Subjects must have adequate bone marrow, renal and hepatic function and coagulation
* Subjects must have normal or clinically insignificant ECG at screening
* Women of reproductive potential must have a negative serum pregnancy test obtained within 3 days before the start of anetumab ravtansine
* Women of childbearing potential and fertile men must agree to use adequate contraception when sexually active. This applies from the time period between signing of the informed consent until at least 6 months after the last administration of the last study drug. Male patients with a female partner of childbearing potential must use a condom and ensure that an additional form of contraception is also used during treatment and until 6 months after last study drug administration.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, superficial noninvasive bladder tumors or any previous cancer curatively treated ≥ 3 years before the start of anetumab ravtansine
* New or progressive brain or meningeal or spinal metastases
* Corneal epitheliopathy or any eye disorder that may predispose the subjects to drug-induced corneal epitheliopathy, or may interfere with diagnosis of treatment-emergent corneal epitheliopathy at the ophthalmologist's or the investigator's discretion
* History or current evidence of

  * biliary cirrhosis
  * malignant biliary obstruction unless the bile flow to the gastrointestinal tract is maintained by a fully operational biliary stent
  * CTCAE (Common Terminology Criteria for Adverse Events) Grade ≥2 bleeding disorder within 4 weeks before the start of anetumab ravtansine
  * uncontrolled cardiovascular disease or uncontrolled hypertension
  * Long QT Syndrome
  * HIV infection
  * Hepatitis B or C infection
* Had a major surgery or significant trauma within 4 weeks before the start of anetumab ravtansine
* Had solid organ or bone marrow transplantation
* Have LVEF (left ventricular ejection fraction) <50% at screening
* Have QTc >450 ms or heart rate ≥100 bpm or ≤45 bpm at screening
* Poor CYP2D6 metabolizers based on the screening test for genetic polymorphisms in CYP2D6 metabolizing capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
PR interval duration | Up to 2 months per patient
  ECG evaluation
QRS interval duration | Up to 2 months per patient
  ECG evaluation
QT interval duration | Up to 2 months per patient
  ECG evaluation
Abnormal T/U waves | Up to 2 months per patient
  ECG evaluation
Heart rate | Up to 2 months per patient
  ECG evaluation
Cycle 1+2 AUC (area under the plasma concentration vs. time curve from zero to infinity after single (first) dose) of BAY94-9343 analytes | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 10h, 24h, 48h, 168h, 336h, 480h and 504h after each dose during first 42 days of the study
Cycle 1+2 AUC(0-tlast) (AUC from time zero to the last data point > LLOQ [lower limit of quantification]) of BAY94-9343 analytes | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 10h, 24h, 48h, 168h, 336h, 480h and 504h after each dose during first 42 days of the study
Cycle 1+2 Cmax (maximum drug concentration in plasma after the first dose administration) of BAY94-9343 analytes | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 10h, 24h, 48h, 168h, 336h, 480h and 504h after each dose during first 42 days of the study
QTcF (QT interval, corrected for heart rate according to Fridericia's formula) interval duration | Up to 2 months per patient
  ECG evaluation
QTcP (QT interval, corrected for heart rate using a population-specific correction) interval duration | Up to 2 months per patient
  ECG evaluation

SECONDARY OUTCOMES:
Incidence of serious adverse events | Up to 6 months per patient
Incidence of non-serious adverse events | Up to 6 months per patient
Incidence of positive anti-drug antibody titer | Up to 6 months per patient
Incidence of neutralizing antibody titers | Up to 6 months per patient
Cycle 3 Cmax,md (Cmax after multiple-dose administration) of BAY94-9343 analytes | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 168h, 336h and 504h between 43rd and 64th days of the study
Cycle 3 AUC(0-tlast)md (AUC(0-tlast) after multiple-dose administration) of BAY94-9343 analytes | At pre-dose, 0.5h, 1h, 1.5h, 2h, 3h, 5h, 8h, 168h, 336h and 504h between 43rd and 64th days of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- United States (5):
  - UCLA-Santa Monica Medical Center, Santa Monica, California
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mary Crowley Medical Research Center, Dallas, Texas
- Australia (2):
  - Blacktown Cancer & Haematology Centre, Blacktown, New South Wales
  - Epworth HealthCare, Richmond, Victoria
- Belgium (2):
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
- France (3):
  - Hôpital Henri Mondor, Créteil
  - Centre Georges Francois Leclerc Dijon, Dijon
  - Hôpital de la Timone - Marseille, Marseille
- Netherlands (3):
  - Nederlands Kanker Instituut, Amsterdam
  - VUmc, Amsterdam
  - Universitair Medisch Centrum St. Radboud, Nijmegen
- Spain (3):
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz (Clinica de la Concepcion), Madrid
  - Hospital Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/